CLINICAL TRIAL: NCT00835406
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Teva Pharmaceuticals USA and Merck Sharp & Dohme (USA) (Fosamax®) Alendronate Sodium Tablets Administered as a 1 x 70 mg in Healthy Adult Males Under Fasting Conditions
Brief Title: Alendronate Sodium 70 mg Tablet Versus Fosamax® Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 00161
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-06-11 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate Sodium First (Experimental): 70 mg Alendronate Sodium Tablets test product dosed in first period followed by 70 mg Fosamax® Tablets reference product dosed in second period
  Interventions: Drug: Alendronate Sodium Tablets 70mg
- Fosamax® First (Active Comparator): 70 mg Fosamax® Tablets reference product dosed in first period followed by 70 mg Alendronate Sodium Tablets test product dosed in second period.
  Interventions: Drug: Fosamax® Tablets 70mg

INTERVENTIONS:
Drug: Alendronate Sodium Tablets 70mg — 1 x 70mg, single dose fasting
  Arms: Alendronate Sodium First
Drug: Fosamax® Tablets 70mg — 1 x 70 mg, single dose fasting
  Arms: Fosamax® First

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of alendronate sodium 70 mg tablets (test) versus Fosamax® 70 mg tablets (reference) administered as a single dose of 70 mg under fasting conditions. A review of pharmacokinetic data demonstrates Alendronate Sodium Tablets, 70 mg, manufactured and distributed by TEVA Pharmaceuticals USA are bioequivalent to Fosamax® Tablets, 70 mg, manufactured by Merck Sharp & Dohme, USA.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males, non-smokers, between 18 and 45 years of age.
* Subjects' weight will be within 15% of their ideal body weight based on the Table of "Desirable Weight of Adults", Metropolitan Life Insurance Company, 1983
* Subjects should read, sign, and date an Informed Consent Form prior to any study procedures.
* Subjects must complete all screening procedures within 28 days prior to the administration of study medication.

Exclusion Criteria:

* Clinically significant abnormalities found during medical screening.
* Any history or presence of significant neurological, hepatic, renal, endocrine, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Any clinically significant history of ongoing gastrointestinal problems or problems known to interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. chronic diarrhea, inflammatory bowel diseases).
* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Abnormal laboratory tests judged clinically significant.
* ECG or vital signs abnormalities (clinically significant).
* History of allergic reactions to alendronate or other related drugs (e.g. clodronate, etidronate and pamidronate).
* History of allergic reactions to heparin.
* Any food allergies, intolerances, restrictions, or special diet which in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* Positive urine drug screen at screening or at check-in of period I.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* Use of an investigational drug or participation in an investigational study, within 30 days prior to administration of the study medication.
* Recent donation of plasma (500 mL) within 7 days or recent donation or significant loss of whole blood (450 mL) within 56 days prior to administration of the study medication.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* Recent history of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana, pot) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP), crack) within 1 year of the screening visit.
* Subjects who have used tobacco within 90 days of the start of the study.
* Subjects who have taken prescription medication 14 days preceding administration of study medication or over-the-counter products 7 days preceding administration of study medication, except for topical products without systemic absorption.
* Subjects who have taken any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine).
* Subjects who have undergone clinically significant surgery 4 weeks prior to the administration of the study medication.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2000-06; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Pharm.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Period: First Intervention
Arm/Group | Alendronate Sodium First | Fosamax® First
Started | 70 | 70
Completed | 68 | 69
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: Period: Washout of 7 Days
Arm/Group | Alendronate Sodium First | Fosamax® First
Started | 68 | 69
Completed | 68 | 67
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Period: Second Intervention
Arm/Group | Alendronate Sodium First | Fosamax® First
Started | 68 | 67
Completed | 68 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate Sodium First | Fosamax® First | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 70 | 70 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 70 | 69 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based on Rmax
Description: Rmax = maximum rate of urinary excretion
Time Frame: Urine collected over 36 hour period
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Alendronate Sodium: 70 mg Alendronate Sodium Tablets test product dosed in either period
- Fosamax®: 70 mg Fosamax® Tablets reference product dosed in either period
Arm/Group | Alendronate Sodium | Fosamax®
Number analyzed (Participants) | 135 | 135
ng/mL | 73.96 (40.48) | 73.99 (39.00)
Statistical Analysis 1: Comparison: Alendronate Sodium vs Fosamax®; Test type: Non-Inferiority or Equivalence — ANOVA will be performed on ln-transformed Ae0-36 and Rmax at the α level of 0.05; Ratio of the mean = 97.94, 90% CI [90.96 to 105.45] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: Bioequivalence Based on Ae0-36
Description: Ae0-36 = cumulative urine excretion
Time Frame: Urine collected over 36 hour period
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alendronate Sodium | Fosamax®
Number analyzed (Participants) | 135 | 135
ng/mL | 219.28 (127.25) | 213.44 (118.05)
Statistical Analysis 1: Comparison: Alendronate Sodium vs Fosamax®; Test type: Non-Inferiority or Equivalence — ANOVA will be performed on ln-transformed Ae0-35 and Rmax at the α level of 0.05; Ratio of the mean = 100.36, 90% CI [92.85 to 108.48] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.